CLINICAL TRIAL: NCT01551745
Title: Phase II Trial of Adjuvant Bi-shRNAfurin and GMCSF Augmented Autologous Tumor Cell Vaccine (FANG™) Integrated With Bevacizumab for Patients With Recurrent/Refractory Ovarian Cancer Participating in Study CL-PTL 105
Brief Title: Salvage Ovarian FANG™ Vaccine + Bevacizumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gradalis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-PTL 112
Record Dates: First submitted 2012-03-01; First posted 2012-03-13 (Estimated); Results first posted 2018-05-01 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Stage III Ovarian Cancer; Stage IV Ovarian Cancer
Keywords: Papillary Serous Ovarian Cancer; Endometrioid Ovarian Cancer; Epithelial Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Bevacizumab; Vascular Endothelial Growth Factor A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vigil™ Vaccine (Experimental): Patients will receive 1.0 x 10e7 cells via intradermal injection one day each cycle for a maximum of 12 doses as long as sufficient material is available and subject is clinically stable. Additionally, patients will receive bevacizumab 10 mg/kg intravenously (prior to Vigil™ administration) every 2 weeks (4 weeks=1 cycle).
  Interventions: Biological: Vigil™ Vaccine; Drug: Bevacizumab

INTERVENTIONS:
Biological: Vigil™ Vaccine — Patients meeting eligibility criteria will receive Autologous Vigil™ vaccine will be supplied by Gradalis,Inc. Patients will receive 1.0 x 10e7 cells via intradermal injection one day each cycle for a maximum of 12 doses as long as sufficient material is available and subject is clinically stable. Additionally, patients will receive bevacizumab 10 mg/kg intravenously (prior to Vigil™ administration) every 2 weeks (4 weeks=1 cycle).
  Other Names: bi-shRNA furin and GMCSF Augmented Autologous Tumor Cell Vaccine; formerly known as FANG™
Drug: Bevacizumab — Patients meeting eligibility criteria will receive bevacizumab 10 mg/kg intravenously every 2 weeks.
  Other Names: VEGF

SUMMARY:
This is a Phase II study of Vigil™ autologous tumor cell vaccine integrated with bevacizumab. All patients will have had Vigil™ prepared and stored from initial primary surgical debulking. Patients meeting eligibility criteria will receive Vigil™ 1.0 x 10e7 cells/intradermal injection once every 4 weeks and bevacizumab 10 mg/kg intravenously every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed papillary serous or endometrioid ovarian cancer.
2. Previous randomization to Gradalis, Inc. protocol CL-PTL 105; observation arm (Group B) or patients with vaccine prepared for CLPTL 105 but not otherwise qualifying.
3. Recurrent cisplatinum resistant/refractory disease (defined as the appearance of any measurable or evaluable lesion or as asymptomatic CA-125 levels greater than 100 u/mL at two consecutive measurements with no intervening therapy.
4. Successful manufacturing of 4 vials of Vigil™ vaccine.
5. Recovered from all clinically relevant toxicities related to prior therapies.
6. ECOG PS 0-2 prior to Vigil™ vaccine administration.
7. Normal organ and marrow function as defined below:

   1. Absolute granulocyte count ≥1,500/mm3
   2. Absolute lymphocyte count ≥ 200/mm3
   3. Platelets ≥100,000/mm3
   4. Total bilirubin ≤1.5 x ULN
   5. AST(SGOT)/ALT(SGPT)/alkaline phosphatase ≤2.5 x ULN
   6. Creatinine <1.5 mg/dL
   7. INR < 1.5
8. Baseline blood pressure must be under 140/90
9. Urine protein-to-creatinine ratio < 1.0 mg/dL.
10. Patients must be off all "statin" drugs for ≥ 2 weeks prior to initiation of therapy.
11. Ability to understand and the willingness to sign a written informed protocol specific consent.

Exclusion Criteria:

1. Surgery involving general anesthesia, chemotherapy, radiotherapy, steroid therapy, or immunotherapy within 4 weeks prior to vaccination. Chemotherapy within 3 weeks prior to vaccination. Steroid therapy within 1 week prior to vaccination.
2. Major surgery within 6 weeks or minor surgery within 2 weeks of receiving bevacizumab.
3. Patient must not have received any other investigational agents within 4 weeks prior to study entry.
4. Patients who require parenteral hydration of nutrition and have evidence of partial bowel obstruction or perforation.
5. Patients with history of brain metastases.
6. Patients with compromised pulmonary disease.
7. Short term (<30 days) concurrent systemic steroids ≤ 0.25 mg/kg prednisone per day (maximum 7.5 mg/day) and bronchodilators (inhaled steroids) are permitted; other steroid regimens and/or immunosuppressives are excluded.
8. Prior splenectomy.
9. Prior malignancy (excluding nonmelanoma carcinomas of the skin and carcinoma in situ cervix) unless in remission for ≥ 2 years.
10. Kaposi's Sarcoma.
11. Patients with active bleeding or pathologic conditions that carry high risk of bleeding such as a known bleeding disorder, coagulopathy, or tumor involving major blood vessels.
12. History of Stroke/Transient Ischemic Attack
13. Use of bleeding diathesis
14. Use of anti-coagulants
15. Patients with clinically significant cardiovascular disease including any of the following:

    1. Significant cardiac conduction abnormalities (e.g., PR interval > 0.24 sec or second or third degree AV block.
    2. Uncontrolled hypertension, defined as systolic blood pressure (BP) > 150 mm Hg or diastolic BP > 90 mm Hg.
    3. Myocardial infarction, cardiac arrhythmia, or unstable angina within the past 6 months.
    4. New York Heart Association grade II or greater congestive heart failure.
    5. Serious cardiac arrhythmia requiring medication.
    6. Grade II or greater peripheral vascular disease except episodes of ischemia < 24 hours induration that are managed non-surgically and without permanent deficit
    7. History of cerebrovascular accident within the past 6 months.
    8. No significant traumatic injury within the past 28 days.
16. Uncontrolled infection or psychiatric illness/social situations that would limit compliance with study requirements.
17. Patients with known HIV.
18. Patients with chronic Hepatitis B and C infection.
19. Patients with uncontrolled autoimmune diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minal Barve, MD, Principal Investigator — Mary Crowley Cancer Research Centers
Locations (1):
- Mary Crowley Cancer Research Centers, Dallas, Texas, United States

REFERENCES:
- [Background] Senzer N, Barve M, Kuhn J, Melnyk A, Beitsch P, Lazar M, Lifshitz S, Magee M, Oh J, Mill SW, Bedell C, Higgs C, Kumar P, Yu Y, Norvell F, Phalon C, Taquet N, Rao DD, Wang Z, Jay CM, Pappen BO, Wallraven G, Brunicardi FC, Shanahan DM, Maples PB, Nemunaitis J. Phase I trial of "bi-shRNAi(furin)/GMCSF DNA/autologous tumor cell" vaccine (FANG) in advanced cancer. Mol Ther. 2012 Mar;20(3):679-86. doi: 10.1038/mt.2011.269. Epub 2011 Dec 20. PMID 22186789

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited subjects from CL-PTL-105 who recurred and were either randomized to the control/observation arm (Group B) or screen-failed but had successful manufacturing of Vigil (minimum of 4 doses).
Pre-assignment Details: 5 subjects were enrolled and started Vigil treatment plus Bevacizumab. 2 subjects completed treatment and 3 did not complete treatment due to disease progression (2) and withdrawal of consent (1).
Period: Overall Study
Arm/Group | Vigil™ Vaccine
Started | 5
Completed | 2 ("Completed" means subject had been given all manufactured doses)
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Disease Progression | 2

BASELINE CHARACTERISTICS:
Arm/Group | Vigil™ Vaccine
Number analyzed (Participants) | 5
Age, Customized [Count of Participants; unit: Participants]
  Age: 0-15 Years | 0
  Age: 16-64 Years | 3
  Age: 65 Years and Older | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 5
  Black/African American | 0
  Asian | 0
  Hispanic | 0
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: Time to progression (TTP) following bevacizumab integrated with Vigil vaccine in patients failing standard of care in study CL-PTL 105 or in those not otherwise qualifying after vaccine production. This will be measured from the treatment start date (date of first dose) to either the date the patient is first recorded as having disease recurrence (even if the patient went off treatment because of toxicity), or the date of death if the patient dies due to any causes before progression.
Time Frame: 24 months
Population: 5 subjects were enrolled and started Vigil treatment. 2 subjects completed treatment and 3 did not complete treatment due to disease progression (2) and withdrawal of consent (1). There is no Outcome Measure Data table because Time to Progression (TTP) and Response Rate (RR) were not collected and analyzed. This study was terminated.
Arm/Group | Vigil™ Vaccine
Number analyzed (Participants) | 0

2. Primary Outcome: Response Rate
Description: Response will be evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline.
Time Frame: Up to 12 months
Population: as for outcome 1
Arm/Group | Vigil™ Vaccine
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Alive Subjects
Description: Survival status of patients after treatment was determined by following these patients up to 24 months.
Time Frame: 24 months
Population: 5 subjects were enrolled and started Vigil treatment. 2 subjects completed treatment and 3 did not complete treatment due to disease progression (2) and withdrawal of consent (1). After 24 months, only 1 of the 5 subjects was alive. Statistical analysis was not done. This study was terminated.
Measure: Count of Participants; unit: Participants
Arm/Group | Vigil™ Vaccine
Number analyzed (Participants) | 5
Participants
  Alive Subjects After 24 months | 1
  Dead Subjects After 24 months | 4

4. Secondary Outcome: Enzyme-Linked ImmunoSorbent Spot (ELISPOT)
Description: To determine if subjects will have a positive (defined as >10 ELISPOTS from baseline) immune response to Vigil. Blood was collected to compare ELISPOT results from baseline until 30 days after last dose.
Time Frame: Baseline, End of Treatment (30 days after last dose) up to 12 months
Population: 5 subjects were enrolled and started Vigil treatment. 2 subjects completed treatment and 3 did not complete treatment due to disease progression (2) and withdrawal of consent (1). After 12 months, all 5 subjects had positive ELISPOT response. Statistical analysis was not done. This study was terminated.
Measure: Count of Participants; unit: Participants
Arm/Group | Vigil™ Vaccine
Number analyzed (Participants) | 5
Participants
  ELISPOT-Positive After 12 months | 5
  ELISPOT-Negative After 12 months | 0

ADVERSE EVENTS:
Arm/Group | Vigil™ Vaccine
All-Cause Mortality (participants affected / at risk) | 4/5
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vigil™ Vaccine (N=5)
Acute Cholecystitis (Hepatobiliary disorders) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Intracerebral Hemorrhage (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vigil™ Vaccine (N=5)
Injection Site Reaction (General disorders) | 2 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes